CLINICAL TRIAL: NCT05209451
Title: Increasing Digital Equity and Access Among Rural Patients (IDEA) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christi Patten, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-011617
Record Dates: First submitted 2022-01-10; First posted 2022-01-26 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Smoking Cessation
Keywords: Rural; Smoking; Smoking cessation; Treatment; Intervention; Digital; Literacy; Equity; Inclusion; Community Engagement
MeSH Terms: conditions — Smoking Cessation; Smoking; Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Condition - No additional study intervention (Active Comparator): Subjects will receive a 12-week, digital, evidence-based behavioral health program for smoking cessation delivered through the patient portal and a written guide on existing digital access resources along with any other necessary material.
  Interventions: Behavioral: Digital, evidence-based behavioral health program for smoking cessation
- Loaner Digital Device (Experimental): Subjects will receive a 12-week, digital, evidence-based behavioral health program for smoking cessation delivered through the patient portal and a written guide on existing digital access resources along with any other necessary material. Participants in this group will also receive a loaned Bluetooth enabled iPad with data plan coverage for the study duration.
  Interventions: Behavioral: Digital, evidence-based behavioral health program for smoking cessation; Other: Bluetooth enabled iPad
- Loaner Digital Device + Coaching Support (Experimental): Subjects will receive a 12-week, digital, evidence-based behavioral health program for smoking cessation delivered through the patient portal and a written guide on existing digital access resources along with any other necessary material. Participants in this group will also receive a loaned Bluetooth enabled iPad with data plan coverage for the study duration plus up to six coaching call, 15-20 minutes in duration.
  Interventions: Behavioral: Digital, evidence-based behavioral health program for smoking cessation; Behavioral: Coaching Support

INTERVENTIONS:
Behavioral: Digital, evidence-based behavioral health program for smoking cessation — Remotely delivered, 12-week smoking cessation program delivered through the patient portal. The program will deliver a smoking cessation intervention that links study participants to tailored, interactive and effective evidence-based smoking cessation resources.
Other: Bluetooth enabled iPad — Bluetooth enabled iPad with data plan coverage that provides a personal Wi-Fi (Internet) hot spot for all home devices and allows for up to 64 GB of cellular data.
  Arms: Loaner Digital Device
Behavioral: Coaching Support — Six coaching calls, 15-20 minutes each in duration. The research coach will use motivational interviewing and goal setting to enhance the participant's technology access and use and digital literacy.
  Arms: Loaner Digital Device + Coaching Support

SUMMARY:
The purpose of this research is to learn more about how access to digital resources impacts healthcare and smoking cessation in rural areas of Minnesota, Iowa, and Wisconsin.

Aim 1: Conduct a pragmatic randomized clinical trial and use mixed methods to assess the impact of providing access to technology and/or coaching support on participation in and response to a digital, evidence-based behavioral health program for smoking cessation.

Aim 2: Assess the feasibility and patient experience of providing electronic remuneration and a loaner device with data plan coverage to access the Internet for remote clinical trials participation.

DETAILED DESCRIPTION:
Rural Community Advisory Committee (CAC) The investigators partnered with the Mayo Clinic Community Engagement Program and Center for Health Equity and Community Engaged Research (CHCR) to form a study-specific Community Advisory Committee (CAC) consisting of 13 members. The CAC is comprised of rural patient advocates, community members and other stakeholders (e.g., MCHS clinicians, Minnesota Rural Broadband Coalition representative). The charge of the CAC is to provide advice and co-design all study materials, digital health access interventions, recruitment messaging, and study dissemination materials and strategies. The CAC met three times with the study team virtually by zoom in September, October, and November of 2021, with each meeting about 90 minutes duration. Members provided feedback on the study protocol including the recruitment messaging and materials, as well as the electronic remuneration process, smoking cessation program, and digital access interventions. The protocol and study materials that are included incorporated this feedback. The CAC will meet four times in 2022. Members will receive a $150 honorarium for each meeting attended.

Study Design

This pragmatic trial is a three-arm, randomized, parallel group design with 90 participants. All participants will receive a 12-week, digital, evidence-based behavioral health program for smoking cessation delivered through the patient portal. All participants will also receive a written guide on existing digital access resources and any other necessary materials. Participants will be stratified based on geographic location (MN, IA, WI) and randomized with 1:1:1 allocation to one of three digital health access intervention groups:

1. Control Condition- no additional study intervention (n=30),
2. Loaner Digital Device - participants will be loaned a Bluetooth enabled iPad with data plan coverage for the study duration (n=30),
3. Loaner Digital Device + Coaching Support - participants will receive the same loaner device described for Group 2 plus up to six coaching calls, 15-20 minutes each in duration. The research coach will use motivational interviewing and goal setting to enhance the participant's technology access and use and digital literacy (n=30).

All participants will complete study assessments at baseline, and at 4 and 12-weeks post-randomization. Outcomes will be assessed using mixed methods. The primary outcome is a composite measure of trial engagement derived from measures of online smoking cessation program engagement (e.g., opening portal messages) and study assessment completion. Secondary outcomes are smoking-related treatment response (self-reported smoking abstinence and use of evidence-based cessation treatment). We will also assess patient experience.

Rationale for the design: The study design will allow us to evaluate the impact of providing the iPad device, or written resource materials on accessing the Internet, without the coaching support. The Investigators can therefore draw causal inferences about key components of the intervention that are necessary for success. From our qualitative work assessing patient experience, the Investigators will learn in this project if more intensive, tailored education and support is necessary to address rural culture and contextual factors, consistent with the Digital Health Equity Framework (Crawford et al., 2020). The study design has utility for the Office of Clinical Trials as well as decision makers within the MCHS about the resources needed for rural patients to access clinical trials and health care remotely.

ELIGIBILITY:
Inclusion Criteria:

* A Mayo Clinic Midwest patient (Mayo Clinic Rochester or Mayo Clinic Health System [MCHS]) with a Mayo Clinic number.
* Aged 18 years or older.
* Can read and speak in the English language. Based on 2019 data, 97% of our Rochester and MCHS patients speak English. The study will provide all participants with a smoking cessation program delivered through the Mayo Clinic patient portal. Currently, Mayo Clinic's portal services are not offered in languages other than English.
* Has a Minnesota, Iowa, or Wisconsin address currently or at date of most recent visit to Mayo Clinic.
* Rural resident based on RUCA codes derived from ZIP code of current or last known address.
* Has access to a telephone of any type (e.g., landline, smartphone). Access to a telephone is needed to complete the coaching support intervention and to follow-up with participants if there are issues with accessing the patient portal for the smoking cessation intervention.
* Current smoker defined as one or more cigarettes (even a puff) smoked in the past 30 days (original criteria). This definition allows for enrollment of non-daily and/or light smoking enhancing the generalizability. In addition to cigarettes, cigarillos and cigars are combustible tobacco products and thus relevant as a focus for our study. Thus, the protocol was modified with IRB approval to change this criterion to include other combustible tobacco use. The final criterion was "Current smoker defined as one or more cigarettes, cigarillos, or cigars (even a puff) smoked in the past 30 days." To enhance the generalizability of our findings, we will enroll participants using other tobacco/nicotine products if cigarette, cigarillo or cigar smoking is the primary product used
* For past 3 months not enrolled in a program or use of cessation pharmacotherapy (original criterion). The protocol was modified with IRB approval to allow for ad hoc use to enhance generalizability. The final criterion was "For past 3 months not enrolled in a program or use of cessation pharmacotherapy other than ad hoc use, for example used nicotine gum or lozenge once or twice."
* Willing to make a quit smoking attempt.
* Has a patient portal account, or is willing to create a patient portal account.
* Has an email address to provide to study staff, or is willing to create an email address.
* Has digital access barriers defined by one or more of the following:

  1. based on participant ZIP code from current or last known address geocoded census block group indicates area of poor BB internet coverage; (b) no existing Mayo Clinic patient portal account or (c) has a Mayo Clinic patient portal account but has not used it in the past 5 years; (d) self-reports having no access to broadband (high speed) internet connection for personal use; and/or (e) self-reports low digital literacy defined with the screening question "How comfortable are you using technology to manage your health care remotely? For example, using patient online services (i.e., patient portal) to schedule appointments, check for test results, or send a message to your provider?" (included: not at all or a little comfortable).

Exclusion Criteria:

* Anyone not meeting all inclusion criteria will be excluded.
* Has participated in a behavioral smoking cessation program in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Trial engagement | 12 weeks
  Composite measure of assessment completion and use of online cessation program

SECONDARY OUTCOMES:
Smoking abstinence | 4 and 12 weeks
  Self-reported smoking abstinence
Use of evidence-based smoking cessation treatment | 4 and 12 weeks
  Self-reported use of any cessation treatment
Patient experience | 12 weeks
  Qualitative interviews of participants' experience with the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Christi Patten, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Kelpin S, Brockman TA, Decker PA, Young A, Boehmer K, Nguyen A, Kamath C, St Sauver J, Sinicrope PS, Sharma P, McCoy R, Allen S, Huang M, Pritchett J, Esterov D, Lampman M, Petersen C, Cheville A, Patten CA. Increasing digital equity to promote online smoking cessation program engagement among rural adults: a randomized controlled pilot trial. Commun Med (Lond). 2024 Oct 8;4(1):194. doi: 10.1038/s43856-024-00624-6. PMID 39375517
- [Derived] Patten CA, Koller KR, King DK, Prochaska JJ, Sinicrope PS, McDonell MG, Decker PA, Lee FR, Fosi JK, Young AM, Sabaque CV, Brown AR, Borah BJ, Thomas TK. Aniqsaaq (To Breathe): Study protocol to develop and evaluate an Alaska Native family-based financial incentive intervention for smoking cessation. Contemp Clin Trials Commun. 2023 Apr 3;33:101129. doi: 10.1016/j.conctc.2023.101129. eCollection 2023 Jun. PMID 37091507
- [Derived] Patten C, Brockman T, Kelpin S, Sinicrope P, Boehmer K, St Sauver J, Lampman M, Sharma P, Reinicke N, Huang M, McCoy R, Allen S, Pritchett J, Esterov D, Kamath C, Decker P, Petersen C, Cheville A. Interventions for Increasing Digital Equity and Access (IDEA) among rural patients who smoke: Study protocol for a pragmatic randomized pilot trial. Contemp Clin Trials. 2022 Aug;119:106838. doi: 10.1016/j.cct.2022.106838. Epub 2022 Jun 25. PMID 35760340
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials